CLINICAL TRIAL: NCT02679131
Title: An Open-label, Nonrandomized, Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Belinostat in Patients With Relapsed/Refractory Solid Tumors or Hematological Malignancies Who Have Mild, Moderate, and Severe Renal Impairment
Brief Title: To Evaluate Safety and Pharmacokinetics of Belinostat in Patients Who Have Mild, Moderate and Severe Renal Impairment.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Close out study w/o Cohort D; Severe Impairment (eGFR=15 to <30mL/min/1.73m²)
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-BEL-105
Record Dates: First submitted 2016-01-27; First posted 2016-02-10 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Relapsed/Refractory Solid Tumors/Hematological Malignancies
Keywords: relapsed/refractory solid tumors; beleodaq; renal impairment; belinostat; hematological malignancies
MeSH Terms: conditions — Recurrence; Renal Insufficiency; Hematologic Neoplasms | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Experimental): Normal Renal function, Belinostat IV, Dose A
  Interventions: Drug: Belinostat
- Cohort B (Experimental): Mild Impairment, Belinostat IV, Dose A
  Interventions: Drug: Belinostat
- Cohort C (Experimental): Moderate Impairment, Belinostat IV, Dose B
  Interventions: Drug: Belinostat
- Cohort D (Experimental): Severe Impairment, Belinostat IV, Dose B
  Interventions: Drug: Belinostat

INTERVENTIONS:
Drug: Belinostat — Belinostat will be administered once daily on days 1 to 5 of a 21-day cycle (up to 6 cycles) via 30-min. IV infusion.
  Other Names: Beleodaq

SUMMARY:
A phase I, open-label, nonrandomized study to determine the PK profile of belinostat in patients with relapsed/refractory solid tumors or hematological malignancies in patients with renal impairment. Eligible patients will be assigned to 1 of 4 cohorts (A, B, C or D) based on their level of renal function (normal, mild, moderate, or severe renal impairment) and receive belinostat dose A for normal or mild renal impairment, and dose B for moderate or severe renal impairment.

DETAILED DESCRIPTION:
Study Design:

A phase I, open-label, nonrandomized study to determine safety and pharmacokinetics of belinostat in patients with relapsed/refractory solid tumors or hematological malignancies and to determine the PK profiles in patients with renal impairment. Eligible patients will be assigned to 1 of 4 cohorts (A, B, C or D) based on their level of renal function (normal, mild, moderate, or severe renal impairment) and receive belinostat dose A for normal or mild renal impairment, and dose B for moderate or severe renal impairment.

Enrollment into all cohorts will occur simultaneously rather than sequentially except in the following instance: Before any patient is enrolled in Cohort D, safety will be assessed for at least 1 patient in Cohort C through the end of Cycle 6. If the patient in Cohort C experiences a toxicity that is at least Grade 3 in severity, Cohort D will proceed at a reduced starting dose.

Belinostat will be administered via a 30-minute intravenous (IV) infusion once daily on Days 1 to 5 of a 21-day cycle (for up to 6 cycles). Clinical safety will be monitored in each patient, and up to two dose reductions from the starting dose (not less than 250mg/m^2) is allowed based on pre-defined criteria.

If a patient cannot tolerate the reduced dose due to Grade 3 or 4 toxicity, belinostat administration must be discontinued. Dose escalation is not allowed. Blood samples for PK analysis will be collected from Day 1 to Day 3, and urine samples for PK analysis will be collected from Day 1 to Day 4.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is diagnosed with advanced solid tumors or advanced hematological malignancy that is relapsed/refractory, for which no standard salvage therapy exists.
2. Patient must have received at least 1 prior therapy for the current malignancy and has recovered from any toxicity of the prior therapy at screening.
3. Patient has either normal or impaired renal functions.
4. Patient has adequate hematological and hepatic functions.

Exclusion Criteria:

1. Patient has acute or progressive renal impairment related to disease or any other cause (eg, toxicity, obstructive uropathy due to retroperitoneal disease, proteinuria, nephrotic syndrome), or requires dialysis.
2. Patient has acute HBV or HCV
3. Patient has known human immunodeficiency virus (HIV) positive diagnosis.
4. Patient has had previous exposure to belinostat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Establish pharmacokinetic (PK) profile of belinostat from Area under the Curve (AUC) parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Area under the plasma drug concentration vs. time curve (AUC) at time 0 to tn will be determined based on specified time points of plasma sample collection from Day 1 to Day 3 of belinostat administration
Establish pharmacokinetic (PK) profile of belinostat from Volume of Distribution (Vdss) parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Volume of Distribution (Vdss) proportionality of drug confined to the plasma vs proportion distributed to other tissues will be determined based on total dose of the drug over specified time points of plasma sample collection from Day 1 to Day 3 of belinostat administration
Establish pharmacokinetic (PK) profile of belinostat from Total Body Clearance (CLtot) parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Total Body Clearance (CLtot) of the drug will be determined by the specified time points of in the Urine PK sample collection from Day 1 to Day 4 of belinostat administration.
Establish pharmacokinetic (PK) profile of belinostat from Fraction Excreted (Fe) Unchanged parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Fraction of the drug that is excreted unchanged (Fe) in the urine will be determined by dividing renal clearance over the total renal clearance based on Urine PK samples collection from specified time points in Day 1 to Day 4 of belinostat administration.
Establish pharmacokinetic (PK) profile of belinostat from Non Renal Clearance (CLnonren) parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Non renal clearance (CLnonren) of the drug will be determined by total clearance minus renal clearance based on Urine PK sample collections from specified time points in Day 1 to Day 4 of belinostat administration
Establish pharmacokinetic (PK) profile of belinostat from peak concentration (Cmax) parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Peak Concentration (Cmax) rate of absorption will be determined as the highest observed concentration in a concentration-time profile of Plasma PK sample collection from Day 1 to Day 3 of belinostat administration
Establish pharmacokinetic (PK) profile of belinostat half-life (t1/2) parameters in patients based on renal impairments in cohorts A,B, C, & D | 26 weeks
  Half-life (t1/2 ) of the drug will be determined by by volume of distribution (Vdss) over clearance (Cl) based on specified time points of plasma sample collection from Day 1 to Day 3 of belinostat administration

SECONDARY OUTCOMES:
Number and percentage of patients with any TEAEs by SOC (System Organ Class) and Preferred Term (PT) | First dose of study drug until 30 days after last dose
  safety analysis of patients with onset of treatment emergent related events from Grade 1-5 of the most common TEAE: nausea, fatigue,pyrexia, anemia, vomiting, thrombocytopenia, dypsnea, neutropenia and hypokalemia
Number and percentage of patients with any SAEs by SOC (System Organ Class) and Preferred Term (PT) | First dose of study drug until 30 days after last dose
  safety analysis of patients with serious adverse events includes pneumonia, pyrexia, infection,anemia, deep vein thrombosis, blood creatinine increase, multi-organ failure, and pulmonary embolism
Number and percentage of patients with any TEAEs related to belinostat by SOC (System Organ Class) and Preferred Term (PT) | First dose of study drug until 30 days after last dose
  safety analysis of patients with new onset of treatment emergent adverse event related to study drug based on pyrexia, thrombocytopenia and blood creatinine increase
Number and percentage of patients with any TEAEs causing discontinuation of the study by SOC (System Organ Class ) and PT (Preferred Term) | First dose of study drug until 30 days after last dose
  safety analysis of patients who discontinued treatment based on anemia, fatigue, febrile neutropenia, pneumonia, & multi-organ failure

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Khan, MD, Study Director — Acrotech Biopharma Inc.
Locations (2):
- United States (2):
  - Innovative Clinical Research Institute, Whittier, California
  - Gabrail Cancer Center Research, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No